CLINICAL TRIAL: NCT01573910
Title: An Evaluation of the Safety and Efficacy of Moxifloxacin Ophthalmic Solution 0.5% Versus Ofloxacin Ophthalmic Solution 0.3% in the Treatment of Bacterial Conjunctivitis in Chinese Patients
Brief Title: An Evaluation of the Safety and Efficacy of Moxifloxacin Ophthalmic Solution 0.5% ((VIGAMOX®) Versus Ofloxacin Ophthalmic Solution 0.3% in the Treatment of Bacterial Conjunctivitis in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-10-051
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Bacterial Conjunctivitis
Keywords: Bacterial conjunctivitis; Anti-infective; Antibiotics
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Experimental): Moxifloxacin ophthalmic solution, 0.5%, 1 drop instilled 3 times per day (TID) in each eye for 7 days with a test-of-cure (TOC) at Day 9
  Interventions: Drug: Moxifloxacin ophthalmic solution, 0.5%
- Ofloxacin (Active Comparator): Ofloxacin ophthalmic solution, 0.3%, 1 drop instilled 3 times per day (TID) in each eye for 7 days with a test-of-cure (TOC) at Day 9
  Interventions: Drug: Ofloxacin ophthalmic solution, 0.3%

INTERVENTIONS:
Drug: Moxifloxacin ophthalmic solution, 0.5%
  Other Names: VIGAMOX®
  Arms: Moxifloxacin
Drug: Ofloxacin ophthalmic solution, 0.3%
  Other Names: Tarivid® Eye Drops
  Arms: Ofloxacin

SUMMARY:
The purpose of this study is to evaluate Moxifloxacin 0.5% relative to Ofloxacin 0.3% in the treatment of bacterial conjunctivitis in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Chinese.
* Diagnosis of bacterial conjunctivitis based on clinical observation.
* Understand and sign the approved informed consent. Legally authorized representative can provide informed consent for patients less than 18 years old and/or incapable of understanding the informed consent.
* Willing to complete all required study procedures and visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women who are pregnant, lactating, or planning a pregnancy.
* Only 1 sighted eye or vision not correctable to 0.6 logMAR or better in either eye.
* Planned contact lens wear during the course of the study.
* Signs and symptoms of bacterial conjunctivitis for longer than 4 days prior to Screening (Day 1).
* Suspected fungal, viral, or Acanthamoeba infection.
* Any systemic or ocular disease or disorder, complicating factor or structural abnormality that would negatively affect the conduct or outcome of the study.
* History of recent surgery.
* Presence of concomitant systemic viral infection.
* Other protocol-defined exclusion criteria may apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 985 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Yu, Lead CSM, Study Director — Alcon Research
Locations (1):
- Alcon (China) Ophthalmic Product Co., Ltd., Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 16 study centers located in China.
Pre-assignment Details: Of the 985 enrolled, 3 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (982).
Groups:
- Moxifloxacin; Ofloxacin: 1 drop instilled TID in each eye for 7 days with a TOC at Day 9
Period: Overall Study
Arm/Group | Moxifloxacin | Ofloxacin
Started | 489 | 493
Completed | 469 | 476
Not Completed | 20 | 17
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Patient decision unrelated to Advs Event | 11 | 11

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who were administered study medication or potentially used study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin | Ofloxacin | Total
Number analyzed (Participants) | 489 | 493 | 982
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (15.54) | 38.4 (15.83) | 37.9 (15.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 265 | 519
  Male | 235 | 228 | 463

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate
Description: Ocular signs of bacterial conjunctivitis (bulbar conjunctival injection and conjunctival discharge/exudates) were rated by the investigator on a 4-point scale, with 0=normal/absent; 1=mild; 2=moderate, and 3=severe. Clinical cure rate is presented as the percentage of participants for which the sum of the numerical scores for the 2 cardinal ocular signs of bacterial conjunctivitis was 0 at Day 9 TOC/Exit Visit.
Time Frame: Day 9
Population: This analysis population includes all patients who received study medication, had no major protocol deviations, had bacteria present at Day 1 visit, and had baseline and TOC/exit data or early exit data.
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | Ofloxacin
Number analyzed (Participants) | 295 | 291
percentage of participants | 85.4 | 81.4

2. Primary Outcome: Microbiological Success Rate
Description: Microbiological specimen(s) from the affected eye(s) were collected according to a protocol-defined process. Microbiological success rate is presented as the percentage of participants for which the pre-therapy pathogens at Visit 1 (Day 1) were eradicated at Day 9 TOC/Exit Visit.
Time Frame: Day 9
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxifloxacin | Ofloxacin
Number analyzed (Participants) | 295 | 291
percentage of participants | 95.3 | 94.8

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (May 2012 to April 2014). This analysis group includes all patients who were administered or potentially used study medication.
Description: An adverse event was defined as any untoward medical occurrence in a patient who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment.
Arm/Group | Moxifloxacin | Ofloxacin
Serious Adverse Events (participants affected / at risk) | 1/489 | 0/493
Other Adverse Events (participants affected / at risk) | 0/489 | 0/493
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin (N=489) | Ofloxacin (N=493)
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.